CLINICAL TRIAL: NCT04097834
Title: Integrating PrEP Into Family Planning Services at Title X Clinics in the Southeastern US
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-1784; 5U24HD089880 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-09-20 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Self-collected vaginal swabs; Self-collected anal swabs; Self-collected oral swabs; Blood samples; Urine samples; Hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PrEP Prescription at Enrollment
- No PrEP Prescription at Enrollment

SUMMARY:
Pre-exposure Prophylaxis (PrEP) is a daily pill to prevent HIV that, when taken as prescribed, reduces the risk of getting HIV from sexual intercourse or drug use. In the United States, most studies which examine prescribing PrEP have not included young women. PrEP provides a way for women to take control of their HIV prevention and may be a good option for some women.

Family planning clinics are a trusted source of preventative, routine, and symptom-driven gynecological care for adolescent and young adult women (AYAW). Thus, these clinics are a natural setting to provide PrEP services for AYAW. This study will examine how effectively three clinics in Atlanta are able to implement a PrEP program for their eligible female patients as well as follow a cohort of 300 women for six months (150 starting PrEP immediately and 150 electing to not take PrEP, at least initially) to characterize individual, provider, and clinic-level variables and constructs that are associated with PrEP uptake, continuation, and adherence.

Both participant and biological data will be collected to answer the primary research question. Women will provide blood, urine, oral, vaginal, anal, and hair samples at three different time points. These samples will be tested to measure incident sexually transmitted infections and unplanned pregnancies as well as PrEP adherence (for women who initiated PrEP). Ultimately, this data will describe each clinic's effectiveness at providing PrEP services to AYAW.

DETAILED DESCRIPTION:
Planning4PrEP is a mixed hybrid Type 1 effectiveness implementation study of three family planning clinics in Atlanta integrating PrEP into their services and evaluating the multi-level factors associated with PrEP reach, level of adoption, and implementation (e.g., PrEP screening and prescription) within and across these clinics while also evaluating the effect on PrEP uptake, continuation, and adherence over a six-month follow-up period. Variation exists among types of family planning clinics, and this variation could have an impact on how clinics decide to implement, integrate, and even sustain PrEP services. This study will evaluate three family planning clinics as they adopt and sustain PrEP into their routine services to capture details of the implementation process unique to each clinic type, as well as commonalities across the clinics, with the ultimate aim to evaluate the impact of the implementation on the primary outcome (PrEP uptake, adherence, and continuation).

ELIGIBILITY:
Inclusion Criteria:

1. Must be self-identified as born female
2. Must be able to be provide written informed consent
3. Must be able to speak and understand English as determined by staff during recruitment
4. Must be 13-45 years old at time of consent
5. Must have been seen for a patient visit in one of the three implementation clinics during the preceding 60 days and identified as a PrEP candidate based on point-of-care HIV testing and risk assessment

Exclusion Criteria:

1. HIV-infected at the time of screening by self-report or screening laboratory assessment
2. Currently enrolled in an HIV vaccine trial
3. Has any condition that in the opinion of study staff would make participation in the study unsafe or interfere with achieving study objectives
4. Has been on PrEP for 7 or more consecutive days in the past
5. Currently receiving PrEP services at any location outside the 3 implementation clinics
6. Currently participating in another PrEP or candidate PrEP study

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women ages 13-45 years who have been identified as PrEP eligible in one of the 3 enrolling FP clinics comprise the study population. PrEP eligibility will be based on clinic-performed HIV testing and risk assessment. All participants will be either PrEP-naïve (no periods of PrEP use longer than 7 consecutive days) at baseline or recipient of a PrEP prescription within the past 60 days (with no periods of PrEP use longer than 7 consecutive days prior to this prescription).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a PrEP prescription at baseline who initiate PrEP | 6 months post enrollment
  Among participants with a PrEP prescription at baseline, the proportion who initiate PrEP measured via pharmacy prescription fill data, medical chart abstraction, and participant self-report
Proportion of participants with a PrEP prescription at baseline who attend at least one follow-up visit and have at least one documented PrEP prescription refill during each 3-month interval | 6 months post enrollment
  Among participants with a PrEP prescription at baseline, the proportion who continue their PrEP regimen evidenced by pharmacy prescription fill data, medical chart abstraction, and participant self-report
Percentage of participants with a PrEP prescription at baseline who adhere to their PrEP regimen | 6 months post enrollment
  Among participants with a PrEP prescription at baseline, percentage who adhere to PrEP, defined by 3 data sources at each follow-up visit-pharmacologic, self-report, and pharmacy. Pharmacological data will include: average ng/mg tenofovir (TFV) concentration measured via hair sample; percentage of participants with adherence level consistent with 7 doses/week (TFV ng/mL≥ 0.0370 ng/mL); percentage of participants with dried blood spot TFV concentration≥1250 fmol/punch; percentage of participants with urine TFV immunoassay detected. Self-report data will include: percentage of participants reporting no missed doses in the past 7 days; percentage of participants reporting very good or excellent adherence (5 or 6 on a 6-level scale) in the past 30 days; percentage of participants who self-report adherence of ≥90%. Pharmacy fill data will include: percentage of participants with 80% adherence measured by medication possession ratio (the # of dispensed pills/# of days since starting PrEP)

SECONDARY OUTCOMES:
Incidence rate of Neisseria gonorrhea among each participant group | 3- and 6-months post enrollment
  For each participant group (those with and those without a PrEP prescription at baseline) the incidence rate of STIs per total follow-up period will be calculated as the ratio of new STI infections (confirmed via multiplex PCR testing or chart review) to the total amount of person-time in each group
Incidence rate of Chlamydia trachomatis among each participant group | 3- and 6-months post enrollment
  For each participant group (those with and those without a PrEP prescription at baseline) the incidence rate of STIs per total follow-up period will be calculated as the ratio of new STI infections (confirmed via multiplex PCR testing or chart review) to the total amount of person-time in each group
Incidence rate of Trichomonas vaginalis among each participant group | 3- and 6-months post enrollment
  For each participant group (those with and those without a PrEP prescription at baseline) the incidence rate of STIs per total follow-up period will be calculated as the ratio of new STI infections (confirmed via multiplex PCR testing or chart review) to the total amount of person-time in each group
Incidence rate of unintended pregnancy among each participant group | 3- and 6-months post enrollment
  For each participant group (those with and those without a PrEP prescription at baseline) the incidence rate of unintended pregnancies (pregnancies that do not match a participant's self-reported pregnancy intentions) per total follow-up period will be calculated as the ratio of new pregnancies (confirmed via positive urine pregnancy test) to the total amount of person-time in each group
Incidence rate of HIV infection among each participant group | 3- and 6-months post enrollment
  For each participant group (those with and those without a PrEP prescription at baseline) the incidence rate of HIV infection per total follow-up period will be calculated as the ratio of new HIV infections (defined as a positive HIV test based on an FDA-approved HIV test with confirmatory negative testing of samples collected at baseline) to the total amount of person-time in each group
Proportion of participants among each participant group reporting contraception use | Enrollment and 3- and 6-months post enrollment
  For each participant group (those with and those without a PrEP prescription at baseline), contraception use will be calculated as the percentage of participants who self-report use of a CDC-defined Tier 1 or Tier 2 contraception method
Proportion of participants among each participant group reporting current contraception type | Enrollment and 3- and 6-months post enrollment
  For each participant group (those with and those without a PrEP prescription at baseline), contraception type will be determined as the self-reported current contraception type used
Proportion of participants adherent to current contraceptive method measured among each participant group | Enrollment and 3- and 6-months post enrollment
  Proportion of participants adherent to current contraceptive method measured among each participant group via self-report
Proportion of participants who are clinically-indicated to initiate PrEP | 3- and 6-months post enrollment
  Among all participants, the proportion of participants whose current clinical and behavioral profile indicate, per CDC clinical practice guidelines, they could begin PrEP, measured via STI testing, medical chart review, and self-report
Proportion of participants who indicate interest in initiating PrEP | Enrollment and 3- and 6-months post enrollment
  Among all participants, the proportion of participants who report interest in beginning PrEP via interviewer-administered questionnaire and self-report
Proportion of all participants who initiate PrEP | Enrollment and 3- and 6-months post enrollment
  Among all participants, the proportion of participants with a PrEP-prescription, pharmacy-confirmed fill of their PrEP prescription, and who self-report initiating PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Sales, PhD, Principal Investigator — Emory University; Anandi N Sheth, MD, MSc, Principal Investigator — Emory University; Matthew A Psioda, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study dataset will be submitted and made publicly available to the NICHD's Data and Specimen Hub (DASH) after completion of the study in accordance with the NICHD DASH Data Archive Policy.
Time Frame: De-identified data will become available on the DASH hub no later than the acceptance for publication of the main findings from the final dataset
Access Criteria: De-identified dataset will be publicly available on the DASH hub.

REFERENCES:
- [Background] Koss CA, Hosek SG, Bacchetti P, Anderson PL, Liu AY, Horng H, Benet LZ, Kuncze K, Louie A, Saberi P, Wilson CM, Gandhi M. Comparison of Measures of Adherence to Human Immunodeficiency Virus Preexposure Prophylaxis Among Adolescent and Young Men Who Have Sex With Men in the United States. Clin Infect Dis. 2018 Jan 6;66(2):213-219. doi: 10.1093/cid/cix755. PMID 29020194
- [Background] Liu AY, Yang Q, Huang Y, Bacchetti P, Anderson PL, Jin C, Goggin K, Stojanovski K, Grant R, Buchbinder SP, Greenblatt RM, Gandhi M. Strong relationship between oral dose and tenofovir hair levels in a randomized trial: hair as a potential adherence measure for pre-exposure prophylaxis (PrEP). PLoS One. 2014 Jan 8;9(1):e83736. doi: 10.1371/journal.pone.0083736. eCollection 2014. PMID 24421901
- [Background] Wilson IB, Lee Y, Michaud J, Fowler FJ Jr, Rogers WH. Validation of a New Three-Item Self-Report Measure for Medication Adherence. AIDS Behav. 2016 Nov;20(11):2700-2708. doi: 10.1007/s10461-016-1406-x. PMID 27098408
- [Background] Amico KR, Marcus JL, McMahan V, Liu A, Koester KA, Goicochea P, Anderson PL, Glidden D, Guanira J, Grant R. Study product adherence measurement in the iPrEx placebo-controlled trial: concordance with drug detection. J Acquir Immune Defic Syndr. 2014 Aug 15;66(5):530-7. doi: 10.1097/QAI.0000000000000216. PMID 24853306
- [Background] Haberer JE, Bangsberg DR, Baeten JM, Curran K, Koechlin F, Amico KR, Anderson P, Mugo N, Venter F, Goicochea P, Caceres C, O'Reilly K. Defining success with HIV pre-exposure prophylaxis: a prevention-effective adherence paradigm. AIDS. 2015 Jul 17;29(11):1277-85. doi: 10.1097/QAD.0000000000000647. PMID 26103095
- [Derived] Sheth AN, Hussen SA, Escoffery C, Haddad LB, Powell L, Brown N, Filipowicz TR, McCumber M, Sanchez M, Renshaw L, Psioda MA, Sales JM. Pre-Exposure Prophylaxis Integration Into Family Planning Services at Title X Clinics in the Southeastern United States: Protocol for a Mixed Methods Hybrid Type I Effectiveness Implementation Study (Phase 2 ATN 155). JMIR Res Protoc. 2020 Sep 25;9(9):e18784. doi: 10.2196/18784. PMID 32975528